CLINICAL TRIAL: NCT02141490
Title: Evaluation of Ferumoxytol Enhanced MRI for the Detection of Lymph Node Metastases in Genitourinary (Prostate, Bladder and Kidney) Cancers
Brief Title: Study of Ferumoxytol Enhanced MRI for Detecting Lymph Node Metastases in Prostate, Bladder, and Kidney Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ismail B. Turkbey, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140107; 14-C-0107
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer; Bladder Cancer; Kidney Cancer
Keywords: Lymph Node; Biopsy; Metastatic Nodes; Imaging Agent
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms | interventions — Ferrosoferric Oxide; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferumoxytol + Magnetic Resonance Imaging (MRI) (Experimental): Ferumoxytol +MRI
  Interventions: Drug: Ferumoxytol; Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Ferumoxytol — 7.5mg/kg intravenous (IV) infusion
  Other Names: Feraheme
Diagnostic Test: Magnetic Resonance Imaging (MRI) — 3 MRIs: pre-infusion, 24 and 48 hours post-infusion

SUMMARY:
Background:

People with prostate, bladder, or kidney cancer often have their cancer spread (metastasize) to lymph nodes. It is important for your doctor to know if this has occurred but currently it can be hard to determine if this has occurred on standard imaging studies like computed tomography (CT) or magnetic resonance imaging (MRI). This study uses an agent called Ferumoxytol to identify lymph nodes that might be involved by cancer.

Objective:

- To see how well Ferumoxytol can detect lymph node metastases in patients with prostate, bladder, or kidney cancer.

Eligibility:

-Adults over age 18 with prostate, bladder, or kidney cancer with lymph node involvement.

Design:

* Participants will be screened with a medical history.
* Participants will have blood drawn and a physical exam. Their vital signs will be measured. They will answer questions about their health and current medications.
* Participants should not have a history of iron overload or have an allergy to Ferumoxytol.
* Participants will have a magnetic resonance imaging (MRI) scan. The scanner is a metal cylinder with a strong magnetic field. Participants will lie on a table that slides in and out of the scanner. They will have a standard sensor, known as a coil, wrapped around their abdomen to improve the scan. This is like a small blanket with wiring inside. Participants will need to lie still on the scanning table for about 1 hour.
* Participants will have an ultrasound. This uses harmless sound waves to provide pictures of organs or tissues inside the body.
* Participants will receive an injection of Ferumoxytol through an intravenous line. A very thin plastic tube will be inserted into a vein in order to inject the agent.
* Participants will have another MRI and ultrasound 24 and 48 hours after injection.
* The study will follow participants medical course for at least 1 year.

DETAILED DESCRIPTION:
Background:

* Conventional imaging modalities (e.g. computed tomography [CT] and magnetic resonance imaging [MRI]) are currently used for the detection of lymph node metastases in many cancer types, including prostate, bladder and kidney cancers, however diagnosis is based on node enlargement which is neither sensitive nor specific (i.e. small nodes harbor metastases, large nodes can be hyperplastic).
* As a consequence, the standard of care is to remove numerous lymph nodes during surgery or to biopsy enlarged nodes to ascertain lymph node status.
* In 2003 Dextran coated ultra small superparamagnetic iron oxide particles (USPIO), also known as Ferumoxtran-10 (Combidex, AMAG Pharmaceuticals, Inc. Lexington, Massachusetts (MA), United States (US)) was shown to localize lymph node metastases with much greater accuracy than unenhanced MRI. Although a large study in prostate cancer was successful, and Food and Drug Administration (FDA) Advisory Panel did not recommend approval and the company abandoned the agent.
* In 2009 Ferumoxytol (Feraheme AMAG Pharmaceuticals, Inc. Lexington, MA, United States (US)) a semi-synthetic carbohydrate coated, magnetic iron oxide preparation similar to ferumoxtran 10 was approved for iron replacement therapy. Like ferumoxtran 10, this compound is taken up by normal lymph nodes and excluded from malignant nodal tissue.
* Results of a recent National Cancer Institute (NCI) trial (11-C-0098) in 15 patients revealed that using the dose of 7.5 mg/kg Fe is safe and yields homogenous and accurate signal changes in benign lymph nodes in comparison with the 4 and 6 mg/kg Fe doses. This dose was further tested in 5 patient's with known or suspected nodal involvement from prostate cancer and in four of five patients positive lymph nodes had a lower signal drop than the benign nodes. The one case in which there was uptake by positive nodes may have been on a vascular basis. This pilot study stimulated interest in a larger study involving a variety of cancer types.

Primary Objective:

-To compare the difference in signal between metastatic and normal nodes in prostate, kidney and bladder cancer patients.

Eligibility

* Subject must be greater than or equal to 18 years old.
* Eastern Cooperative Oncology Group Performance score of 0 to 2.
* There are 3 parallel arms in this study. All patients must have evidence of lymph node involvement (with a short axis diameter greater than or equal to 1.5 cm).
* In addition:
* Arm 1: Subject must have a documented diagnosis of prostate cancer.
* Arm 2: Subject must have a documented diagnosis of bladder cancer (transitional cell carcinoma).
* Arm 3: Subject must have a documented diagnosis of kidney cancer (all renal cell cancer types).

Design:

* This is a single site 3-arm (arm 1=prostate cancer, arm 2=bladder cancer, arm 3=kidney cancer) study enrolling 50 evaluable patients (30 evaluable in each arm 1, 10 evaluable in arms 2 and 3) with documented prostate, bladder or kidney cancer with evidence of lymph node involvement [with a size of greater than or equal to 1.5 cm measured on conventional imaging (e.g. CT, MRI)].
* All subjects will undergo pre-infusion, 24, 48 hours post-Ferumoxytol infusion (dose of 7.5mg/kg Fe) MRI consisting of T1 weighted (W), T2W and T2*W 3 Tesla MRI.
* Imaging will be correlated with histology of resected or biopsied lymph nodes when available. Occasionally, patients may not undergo biopsy or surgical excision of their lymph nodes. This may occur if their lymph nodes are overtly large and therefore highly likely to represent lymph node involvement. In such cases, patients will be evaluated with clinical follow up which typically occurs every three months in most NCI protocols. If the lesion demonstrates growth or regression based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria on these follow up studies' then the lesion will be considered positive for tumor. If it is stable for at least one year, then it will be considered non-malignant. The MR imaging analysis will be intra-patient.
* Patients will also undergo ultrasound examination of imageable lymph nodes (e.g. inguinal nodes) at pre-infusion and 24, 48 hours post-Ferumoxytol infusion time points. The signal changes at post-infusion ultrasound will be visually evaluated to determine if the uptake of ferumoxytol alters sonographic features.

ELIGIBILITY:
* INCLUSION CRITERIA

2.1.1.1 Subject must be greater than or equal to 18 years old.

2.1.1.2 Diagnosis

* Arm 1: Subject must have a documented diagnosis of prostate cancer with evidence of lymph node involvement (with a short axis diameter of greater than or equal to 1.5 cm on a conventional computed tomography (CT) or magnetic resonance (MRI) obtained within 8 weeks of the Ferumoxytol imaging procedure)
* Arm 2: Subject must have a documented diagnosis of bladder cancer (transitional cell carcinoma) with evidence of lymph node involvement (with a short axis diameter of greater than or equal to 1.5cm on a conventional CT or MRI obtained within 8 weeks of the Ferumoxytol imaging procedure)
* Arm 3: Subject must have a documented diagnosis of kidney cancer (all renal cell cancer types) with evidence of lymph node involvement (with a short axis diameter of greater than or equal to 1.5 cm on a conventional CT or MRI obtained within 8 weeks of the Ferumoxytol imaging procedure)

2.1.1.3 Subject must have Eastern Cooperative Oncology Group Performance score greater than or equal to 2.

2.1.1.4 Ability to provide informed consent. All subjects must sign an informed consent form indicating their understanding of the investigational nature and risks of the study before any protocol-related studies are performed.

2.1.EXCLUSION CRITERIA

2.1.2.1 Subjects with known hypersensitivity and allergy to iron.

2.1.2.2 Subjects with evidence of iron overload with a pre-study ferritin level greater than 370 ng/ml and percent saturation of transferrin level greater than 40%. Patients with lab values above these limits may be included in the study if documented hematology consultation rules out hemochromatosis, idiopathic or iatrogenic iron overload.

2.1.2.3 Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.

2.1.2.4 Subjects with severe claustrophobia unresponsive to oral anxiolytics.

2.1.2.5 Subjects with contraindications to MRI.

2.1.2.6 Subjects weighing >136 kg (weight limit for scanner table).

2.1.2.7 Subjects with any type of pacemaker, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI.

2.1.2.8 Subjects with abnormal liver function tests suggesting liver dysfunction (aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) greater than or equal to 3 x of the upper limits of normal; total bilirubin greater than or equal to 2 x the upper limits of normal or >3.0 mg/dl in patients with Gilbert's syndrome).

2.1.2.9 Subjects with other medical conditions deemed by the principal investigator (or associates) to make the subject ineligible for protocol procedures.

2.1.2.10 Women who are pregnant or breast-feeding. The effects of ferumoxytol on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 1 day after study related imaging is completed. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

2.1.3 Inclusion of Women and Minorities.

Members of all races and ethnic groups are eligible for this trial. Women are excluded from arm 1 of this trial as prostate cancer does not occur in females.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismail B Turkbey, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birkhauser FD, Studer UE, Froehlich JM, Triantafyllou M, Bains LJ, Petralia G, Vermathen P, Fleischmann A, Thoeny HC. Combined ultrasmall superparamagnetic particles of iron oxide-enhanced and diffusion-weighted magnetic resonance imaging facilitates detection of metastases in normal-sized pelvic lymph nodes of patients with bladder and prostate cancer. Eur Urol. 2013 Dec;64(6):953-60. doi: 10.1016/j.eururo.2013.07.032. Epub 2013 Jul 30. PMID 23916692
- [Background] Blom JH, van Poppel H, Marechal JM, Jacqmin D, Schroder FH, de Prijck L, Sylvester R; EORTC Genitourinary Tract Cancer Group. Radical nephrectomy with and without lymph-node dissection: final results of European Organization for Research and Treatment of Cancer (EORTC) randomized phase 3 trial 30881. Eur Urol. 2009 Jan;55(1):28-34. doi: 10.1016/j.eururo.2008.09.052. Epub 2008 Oct 1. PMID 18848382
- [Background] Crispen PL, Breau RH, Allmer C, Lohse CM, Cheville JC, Leibovich BC, Blute ML. Lymph node dissection at the time of radical nephrectomy for high-risk clear cell renal cell carcinoma: indications and recommendations for surgical templates. Eur Urol. 2011 Jan;59(1):18-23. doi: 10.1016/j.eururo.2010.08.042. Epub 2010 Sep 15. PMID 20933322
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0107.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Prostate Cancer; Bladder Cancer; Kidney Cancer: Ferumoxytol + Magnetic Resonance Imaging (MRI)
  Ferumoxytol: 7.5mg/kg intravenous (IV) infusion
  Magnetic Resonance Imaging (MRI): 3 MRIs: pre-infusion, 24 and 48 hours post-infusion
Period: Overall Study
Arm/Group | Prostate Cancer | Bladder Cancer | Kidney Cancer
Started | 34 | 6 | 3
Completed | 30 | 6 | 3
Not Completed | 4 | 0 | 0
Not completed — Screening failures | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prostate Cancer | Bladder Cancer | Kidney Cancer | Total
Number analyzed (Participants) | 34 | 6 | 3 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 3 | 3 | 18
  >=65 years | 22 | 3 | 0 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (6.65) | 66.8 (10.25) | 44.3 (9.45) | 64.2 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2
  Male | 34 | 6 | 1 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 6 | 3 | 42
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 0 | 1 | 7
  White | 27 | 6 | 2 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 6 | 3 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change (From Baseline to 24 Hours) Between Metastatic and Benign Nodes
Description: Visible nodes were quantified with manually contoured regions of interest on axial T2*W MRI to obtain the mean signal intensity (SInode). The SI of the visible lymph node was normalized using the mean SI of the adjacent muscle tissue on the same slice (SImuscle). The following equation was used to obtain the normalized SI from the lymph node (SInormal): SInormal=SInode/SImuscle. The calculation formula was 100% * ((SInormal(24hrs)- SInormal(baseline))/ SInormal(baseline)).This image processing method was performed at baseline, 24-hours post-injection MRI studies to define the SI change differences between benign and malignant lymph nodes from baseline to 24 hours post injection.
Time Frame: Baseline and 24 hours
Population: Results are available for 39/43 subjects because 4 were screen failures.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Groups:
- All Participants: Due to low accrual in the bladder and renal arms, all three diseases (Prostate Cancer, Bladder Cancer and Kidney Cancer) were combined together for analysis.
  Ferumoxytol + Magnetic Resonance Imaging (MRI)
  Ferumoxytol: 7.5mg/kg intravenous (IV) infusion
  Magnetic Resonance Imaging (MRI): 3 MRIs: pre-infusion, 24 and 48 hours post-infusion
Arm/Group | All Participants
Number analyzed (Participants) | 39
Percentage Change
  % change from baseline to 24h in metastatic nodes | -33.6 [-39.2 to -28]
  % change from baseline to 24h in benign nodes | -46.9 [-54.8 to -39]

2. Secondary Outcome: Percentage Change for Imaging (From Baseline to 48 Hours) Between Metastatic and Benign Nodes
Description: Visible nodes were quantified with manually contoured regions of interest on axial T2*W MRI to obtain the mean signal intensity (SInode). The SI of the visible lymph node was normalized using the mean SI of the adjacent muscle tissue on the same slice (SImuscle). The following equation was used to obtain the normalized SI from the lymph node (SInormal): SInormal=SInode/SImuscle. The calculation formula was 100% * ((SInormal(48hrs)- SInormal(baseline))/ SInormal(baseline))). This image processing method was performed at baseline, 48-hours post-injection MRI studies to define the SI change differences between benign and malignant lymph nodes from baseline to 48 hours post-injection.
Time Frame: Baseline to 48 hours post injection
Population: Results are available for 39/43 subjects because 4 were screen failures.
Measure: Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | All Participants
Number analyzed (Participants) | 39
Percent Change
  % change from baseline to 48h in metastatic nodes | -24 [-32.2 to -15.8]
  % change from baseline to 48h in benign nodes | -40 [-51.5 to -28.4]

3. Secondary Outcome: Percent Change in Signal Difference Within Metastatic Nodes in Prostate, Kidney, Bladder Cancer Patients at Ultrasonography
Description: Patients will undergo ultrasound examination of imageable lymph nodes at pre-infusion, 24 hours and 48 hours. The signal changes at post-infusion ultrasound will be visually evaluated to determine if the uptake of ferumoxytol alters sonographic features.
Time Frame: pre-infusion, 24 hours and 48 hours
Population: The analysis for this outcome measure was not done because most of the patients had deeply located lymph nodes and logistically ultrasonography analysis was not possible.
Arm/Group | Prostate Cancer | Bladder Cancer | Kidney Cancer
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse events were assessed from the date treatment consent signed to date off study, approximately 3 years, 3 months, and 11 days on the Prostate Cancer Arm/Group; 2 years, 5 months, and 19 days on the Bladder Cancer Arm/Group, and 1 year, 6 months, and
Population: Results are available for 39/43 subjects because 4 were screen failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Prostate Cancer | Bladder Cancer | Kidney Cancer
Number analyzed (Participants) | 30 | 6 | 3
Participants | 6 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date treatment consent signed to date off study, approximately 3 years, 3 months, and 11 days on the Prostate Cancer Arm/Group; 2 years, 5 months, and 19 days on the Bladder Cancer Arm/Group, and 1 year, 6 months, and 22 days on the Kidney Cancer Arm/Group.
Description: Results are available for 39/45 subjects because 6 were deemed screen failures following enrollment.
Arm/Group | Prostate Cancer | Bladder Cancer | Kidney Cancer
All-Cause Mortality (participants affected / at risk) | 1/30 | 1/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 6/30 | 2/6 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Cancer (N=30) | Bladder Cancer (N=6) | Kidney Cancer (N=3)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, "Warm feeling" (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT02141490/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT02141490/ICF_001.pdf